CLINICAL TRIAL: NCT02968394
Title: Influence of Omalizumab Co-treatment on Honey-bee Venom Immunotherapy Failure Due to Systemic Reactions
Brief Title: Omalizumab Treatment in Venom Immunotherapy With Systemic Reactions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University Clinic of Pulmonary and Allergic Diseases Golnik (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NEVIT
Record Dates: First submitted 2016-11-11; First posted 2016-11-18 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Allergy; Bee Venom; Immunotherapy; Omalizumab
MeSH Terms: conditions — Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NEVIT (Experimental): Co treatment with omalizumab during another attempt of immunotherapy introduction
  Interventions: Drug: omalizumab

INTERVENTIONS:
Drug: omalizumab

SUMMARY:
The purpose of this study is to evaluate if omalizumab co-treatment may allow reintroduction of honey bee venom immunotherapy in patients with immunotherapy treatment failure due to systemic reactions.

DETAILED DESCRIPTION:
Some honey bee venom allergic patients cannot be treated with venom immunotherapy due to systemic reactions during immunotherapy - immunotherapy failure due to systemic reactions. High basophil allergen sensitivity is a risk factor for venom immunotherapy failure due to systemic reactions. Omalizumab decreases basophil sensitivity. Venom immunotherapy failure patients will be co-treated with omalizumab during another attempt of immunotherapy introduction. Patients will be clinically and immunologically followed up after the introduction.

ELIGIBILITY:
Inclusion Criteria:

* severe anaphylactic reaction after honey-bee sting (Mueller grade III or IV) confirmed sensitization to honey-bee venom,
* honey-bee venom immunotherapy treatment failure due to systemic reactions.

Exclusion Criteria:

* systemic mastocytosis,
* pregnancy,
* use of beta-adrenergic blocking agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Number of systemic reactions during ultra rush immunotherapy build up phase and maintenance phase followed by omalizumab co-treatment. | 2 months

SECONDARY OUTCOMES:
Changes in basophil sensitivity during omalizumab co-treatment | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Mitja Košnik, MD, PhD, Study Director — University Clinic of Pulmonary and Allergic Diseases Golnik
Locations (1):
- University Clinic of Pulmonary and Allergic Diseases Golnik, Golnik, Slovenia